CLINICAL TRIAL: NCT04491344
Title: Extended Geno- and Phenotyping of Overweight and Obese Children and Adolescents
Brief Title: Leipzig Childhood Obesity Study
Status: Recruiting | Type: Observational
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Antje Koerner, Prof. Dr. med., Prof. Dr. med., University of Leipzig
Other Study IDs: ADI cohort Leipzig
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Childhood Obesity
Keywords: Single nucleotide polymorphisms; Obesity; Insulin resistance; Metabolic syndrome; Oral glucose tolerance test
MeSH Terms: conditions — Pediatric Obesity; Obesity; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * serum samples from oral glucose tolerance testing
  * blood samples for DNA analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Children with overweight and obesity: Overweight and obese children and adolescents visiting the adiposity outpatient clinic.
- adults: follow up of patients into adulthood
- control group: matched control group with children, adolescents and aduts without obesity

SUMMARY:
The aim of this study is to identify polymorphisms that make children and adolescents more prone to obesity and metabolic dysfunction, as well as to identify biomarkers that are linked to causes and consequences of obesity.

DETAILED DESCRIPTION:
In order to identify single nucleotide polymorphisms blood and serum samples during oral glucose tolerance testing are routinely obtained from pediatric patients visiting the adiposity outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* all pediatric patients seen in the adiposity outpatient clinic
* informed patient consent

Exclusion Criteria:

* none

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Overweight and obese children and adolescents
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2002-01; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Gene-dependent association with phenotypical traits in overweight and obese children | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Antje Körner, Prof, MD, Principal Investigator — University of Leipzig
Locations (1):
- University Leipzig Medical Center, Department of Women and Child Health, Center for Pediatric Research Leipzig, Leipzig, Saxony, Germany

REFERENCES:
- See also: Link to the pediatric adiposity outpatient clinic — http://kik.uniklinikum-leipzig.de/kikcms.site,postext,ambulante-betreuung,a_id,262.html?PHPSESSID=t7ag2skgnd7cdc2dng21vh2u26
- See also: Link to Prof Antje Körner's Group — http://kik.uniklinikum-leipzig.de/kikcms.site,postext,childhood-obesity-antje-koerner.html?PHPSESSID=oakfosqa62ik082hs9bo6hsah3